CLINICAL TRIAL: NCT01265355
Title: Community Based Prophylaxis for Rotavirus Gastroenteritis in Children by an Anti-rotavirus Protein Based Food Supplement
Brief Title: Community Based Prevention of Rotavirus Gastroenteritis by a Functional Food Supplement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Christian Medical College, Vellore, India (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CMCLB001
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Rotavirus Gastroenteritis
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anti-rotavirus protein (Experimental)
  Interventions: Dietary Supplement: Anti-rotavirus protein
- Maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Anti-rotavirus protein — 11mg ARP In 1 Gm Product Daily For 12 Months, given in orange juice
  Arms: Anti-rotavirus protein
Dietary Supplement: Maltodextrin — Maltodextrin 1 gm daily
  Arms: Maltodextrin

SUMMARY:
Rotavirus is the commonest cause of severe gastroenteritis in young children worldwide. The investigators hypothesize that use of a food based prophylactic will decrease incidence of rotavirus infection in young children in south India, prevent intestinal damage and overall result in lower infection rates and better gut function. This trial will evaluate the efficacy of prevention of rotavirus gastroenteritis when an anti-rotavirus protein or antibody fragments expressed in yeast or placebo are given daily as a food supplement to children between the ages of 6 and 12 months. The children will followed for one year and rates of rotavirus diarrhoea, antibody responses and gut function will be compared between children receiving antibody fragments or placebo.

DETAILED DESCRIPTION:
The study will be carried out in an urban slum area in Vellore, south India. Children between the ages of 6 and 12 months will be recruited for participation in the study. They will be randomized to receive supplementation with ARP or placebo, and will be followed for a period of one year, with weekly home visits and monitoring of all episodes of diarrhoea. In addition, every two weeks, surveillance stool samples will be collected and tested for rotavirus to identify asymptomatic infections by PCR. All episodes of diarrhoea will be investigated intensively for bacterial, viral and parasitic agents of diarrhoea using both conventional and molecular techniques and all cases will be treated appropriately at the study clinic or referral hospital as required. Monthly anthropometric measurements will be carried out to estimate rates of growth and to identify growth faltering. Blood samples will be taken at 4, 8 and 12 months for estimation of anti-rotavirus IgA and IgG antibodies. Studies on intestinal absorption and permeability will be carried out at recruitment, 6 and 12 months by the lactulose:mannitol test (measured by HPLC detection of sugars). All rotavirus strains obtained will be characterized by genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Healthy child aged 6 to 12 months, families resident in the study area, willing to participate and available for follow up for a period of one year
* Normal birth weight (> 2.5 kg), child exclusively breast fed for at least four months

Exclusion Criteria:

* Families not available for a follow up period of one year
* Children with any atopic conditions
* Children with gross congenital anomalies including cardiovascular, renal or hepatic disease
* Children with syndromic or serological evidence of HIV infection

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence of rotavirus gastroenteritis | One year after recruitment

SECONDARY OUTCOMES:
IgA And IgG Antibody Response To Rotavirus | At 4, 8 And 12 Months after recruitment
Weight For Height Z Score | At 6 and 12 months after recruitment
Intestinal Function by lactulose:mannitol | at 3, 6, 9 and 12 months
Characterization of strains causing rotavirus gastroenteritis | Over 12 months
Incidence of adverse events | Over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gagandeep Kang, MD, Principal Investigator — Christian Medical College, Vellore, India; Uma Raman, MDS, Study Director — Christian Medical College, Vellore, India
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India